CLINICAL TRIAL: NCT04005391
Title: Home-based Delivery of the Contraceptive Implant in Postpartum Guatemalan Women: a Cluster-randomized Trial
Brief Title: Home-based Delivery of the Contraceptive Implant in Postpartum Guatemalan Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 17-1314; 5K12HD001271 (NIH)
Record Dates: First submitted 2019-06-26; First posted 2019-07-02 (Actual); Results first posted 2020-11-24 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Postpartum
Keywords: postpartum contraception; long-acting reversible contraceptives; implant; nursing; community programming; cluster-randomized trial
MeSH Terms: interventions — Condoms; Medroxyprogesterone Acetate; Levonorgestrel

STUDY DESIGN:
Intervention Model Description: Superiority trial to see if home-based postpartum contraceptive delivery, including a long-acting reversible contraceptive, the contraceptive implant, increases uptake of a highly effective method of postpartum contraception (the implant).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Postpartum Contraceptives offered to Intervention Clusters (Experimental): Women will have postpartum contraceptive options (condoms "vive amor", birth control pills "segura plus", injectable "cyclofem", contraceptive implant "jadelle") offered to them at their routine forty day postpartum visit after routine care is provided, first.
  Interventions: Other: Offer of Participant's Choice of Contraception Method
- Routine Care offered to Control Clusters (No Intervention): Women will receive routine postpartum care

INTERVENTIONS:
Other: Offer of Participant's Choice of Contraception Method — Women will be offered a range of contraceptive options (condoms, contraceptive pills, medroxyprogesterone acetate injection, levonorgestrel implant) to choose from; they can decline to start a contraceptive method
  Other Names: condoms; contraceptive pills; medroxyprogesterone acetate injection; levonorgestrel implant
  Arms: Postpartum Contraceptives offered to Intervention Clusters

SUMMARY:
Abstract

Background: Postpartum contraception is important to prevent unintended and closely spaced pregnancies following childbirth.

Methods: This study is a cluster-randomized trial of communities in rural Guatemala where women receive ante- and postnatal care through a community-based nursing program. When nurses visit women for their postpartum visit in the intervention clusters, instead of providing only routine care that includes postpartum contraceptive education and counseling, the nurses will also bring a range of barrier, short-acting, and long-acting contraceptives that will be offered and administered in the home setting, after routine clinical care is provided.

Discussion: A barrier to postpartum contraception is access to medications and devices. The study removes some access barriers (distance, time, cost) by providing contraception in the home. The community nurses were trained to place implants, which are a type of long-acting reversible contraceptive method that was previously only available in the closest town, which is about an hour away by vehicle. Therefore, the study examines how home-based delivery of routinely available contraceptives and the less routinely available implant may be associated with increased uptake of postpartum contraception within three months of childbirth. The potential implications of this study include: nurses may be able to be trained to safely provide contraceptives, including place implants, in the home setting, and provision of home-based contraception may be an effective way of delivering an evidence-based intervention for preventing unintended and closely spaced pregnancies in the postpartum period.

DETAILED DESCRIPTION:
Background and Rationale: Postpartum contraception is important to prevent unintended and closely spaced pregnancies following childbirth as well as to avoid future pregnancy in mothers who have achieved their desired family size. Proper pregnancy spacing can prevent maternal and perinatal morbidity and mortality. Globally, there is significant unmet need for postpartum contraception.

Historically, in the community of interest, which is in the rural Southwest corner of Guatemala bordering Mexico, a large majority (88%) of a convenience sample of women in the community-based care program self-reported postpartum contraceptive use. However, 72% of these women were using injectable contraceptives, which are considered short-acting, and are less effective at preventing unintended and closely spaced pregnancies; the second most common method was sterilization (21%). For the remaining women who did not seek sterilization or injectable contraceptives, 0.5% of them reportedly used contraceptive pills, 0.5% condoms, 0.5% lactational amenorrhea, and 1.6% reportedly relied on natural family planning. Less than 4% of women were using long-acting reversible contraceptives (intrauterine devices or implants), which are more effective at preventing unintended and closely spaced pregnancies than injectables. The providers in the community had not been trained in implant and intrauterine device placement, so the closest place to have a device placed was the most proximate town to the communities, which is an hour away by vehicle. Additional barriers discovered through qualitative research in the study communities found that barriers to family planning use historically included knowledge, access to methods, fear of adverse events, and a woman garnering her partner's approval. Community women's ideas for future educational programming included teaching about how birth control methods work, how to talk to partners about birth spacing, and myth debunking, and they requested the location and time of teaching to occur at peripartum and pediatric visits.

Therefore, based on this preliminary data, the prospective research question is: if community-based nurses are trained to place contraceptive implants, and they offer women placement in the home at their postpartum visit (among other routinely available contraceptive methods), will the ability to provide this service increase the uptake of contraceptive implants in our communities of interest?

Specific Objectives or Hypotheses: The specific objective of the study is to observe in this population where use of postpartum contraception is historically common among women, does home delivery of the contraceptive implant increase utilization of the device above the baseline rate of 3.2%. The investigators hypothesize, based on published data from other settings, that if women receive proper counseling about all contraceptive methods, uptake of long-acting reversible contraceptives, which in this study includes only the contraceptive implant, is about 50%.

The secondary objectives are to observe if the home-based contraceptive delivery intervention featured in this study is associated with overall increased contraceptive uptake, continuation, and satisfaction in the intervention compared to the control clusters. The hypothesis is that with increased uptake of the implant there will be longer continuation rates and more satisfaction in the intervention clusters. The investigators also hypothesize that increased contraceptive uptake, continuation, and satisfaction may be associated with reduced short interval repeat pregnancy rates so the study also aims to survey participants on their pregnancy status at enrollment, and three- and twelve-months after enrollment.

Trial Design: The protocol features an interventional, cluster-randomized, unmasked, parallel group trial design. The eight study communities were randomized in a 1:1 allocation ratio to either the intervention or control arms of the study, and the study is designed on a superiority framework.

Study Setting: The study setting is in the home of women enrolled in the "Madres Sanas" community-based nursing program offered by the Fundación para la Salud Integral de los Guatemaltecos (FSIG). FSIG supports a community-based clinic called the Center for Human Development in a region of Guatemala informally referred to as the Southwest Trifinio. This region is at the intersection of the boundaries of three departments in Guatemala, and as such no single Department takes responsibility for the health of the migrant workers that reside there. The impoverished area has a population of around 25,000 people and experiences poor pregnancy outcomes. This is why the University of Colorado Center for Global Health, in partnership with AgroAmerica, built the Center for Human Development clinic and initiated the community-based maternal and perinatal care programs, called Madres Sanas and Ninos Sanos, respectively.

Madres Sanas is executed by teams of community nurses. The nurse teams are comprised of two nurses, who are responsible for a segment of the communities in the region. There are ten communities in the Madres Sanas program that were combined into eight clusters; our biostastician did this in order to achieve similar cluster sizes, which was determined by the number of births in the communities in 2017. Because our study enrolls women at their final Madres Sanas visit, which is a postpartum visit that occurs about forty days out from delivery, the cluster size was based on delivery volume of the communities. The nurse teams are assigned by the nursing supervisor to their respective communities. They drive auto rickshaws provided by the Center for Human Development out to the communities to conduct their home visits, which include four antenatal visits and two postpartum visits. During the visits the nurses both provide clinical care and collect quality improvement and research data, and as such serve a dual function in their role. As noted, this study takes place at the final Madres Sanas visit, which occurs forty days after delivery. Routine clinical care, including postpartum contraceptive education, culminates at this time, although counseling on postpartum contraception begins at the enrollment visit. After routine clinical care is provided, the nurses offer enrollment in the study.

Interventions: All study activities and procedures begin at the forty-day postpartum visit, which is the sixth and final scheduled visit of the Madres Sanas program. At this visit the community nurses perform routine maternal and neonatal clinical care, which includes amongst other activities, final counseling and education about postpartum contraception. In intervention clusters, nurse teams bring a kit with them to the visit. After the visit they describe the study and offer consent. Once a woman has discussed the risks, benefits, and alternatives with her providers and determines she wishes to participate in the study, she signs the consent form and the nurses offer her condoms, contraceptive pills, a medroxyprogesterone contraceptive injection, or the levonorgestrel implant. The kit is stocked with 10 condoms, one pack of pills, one syringe of medroxyprogesterone, and one implant for each postpartum visit planned for that day. It also contains all the necessary materials to place the implant or administer the injection under sterile conditions, such as alcohol swabs and sterile gloves, etc.

All contraceptives are purchased using study funds and are sourced from a local provider of contraceptive medications and devices. All contraceptives are routinely available and approved for distribution in Guatemala. Because these are routinely available medications and the study does not testing their effectiveness as contraceptives, there are no criteria for discontinuing or modifying allocated interventions for a given trial participant such as changing the drug dosing. Women are, however, screened for contraindications to the contraceptive methods provided using the Medical Eligibility Criteria. The nurses have the eligibility criteria chart in Spanish, laminated, and included in their kit for use during study enrollment. As this is a pragmatic trial, there are no restrictions on care and interventions that are permitted or prohibited during the trial. For example, if a participant did not initiate a contraceptive method and wishes to, she can seek the method in the community. Conversely, if she chose a method and opted for the implant but does not like it, she is free to remove it at any time. The nurses will either remove it in the home setting or advise the woman to present to the Center for Human Development where they can remove it and potentially initiate a new method. The initial contraceptive provided in the study setting is free, but any contraceptives sought or utilized after the study enrollment visit is the woman's responsibility to locate and finance. Study contraceptives are only provided in the home setting by the nurses at the enrollment visit and are not available or offered at any subsequent visit.

Data Collection Methods: Quality improvement data from prior to study initiation was collected from June 2017 - September 2018 by the Madres Sanas community nurses. This database includes antepartum, intrapartum, and postpartum quality improvement data collected by the community nurses during routine antenatal and postnatal care visits. The data is collected on tablets and transmitted through the application REDCap. REDCap (Research Electronic Data Capture) is a secure, HIPAA-compliant web-based application designed for data collection for research studies. It provides an easy-to-use data entry system with data validation, the ability to import data from external sources (Guatemala), automated exports to statistical software, audit trails, branching logic and calculations, and sophisticated tool for building and managing online surveys. As the community nurses have been using this software for years, our study links to the Madres Sanas dataset, but involves separate forms in a separate REDCap database. Just as the nurses prompt women during routine visits and collect general pregnancy outcomes data for our quality improvement database, so will they use REDCap and the same methods to collect enrollment and follow-up on participants and transmit the data to password protected servers at the University of Colorado. There are cluster-specific REDCap forms that are collected on enrollment, at three months, and at twelve months following enrollment.

Statistical Methods: To analyze our primary outcome the investigators are planning a difference in differences analysis of the proportion of women actively using a contraceptive implant three months after enrollment in intervention clusters as compared to control clusters. The investigators plan to provide an unadjusted analysis and an adjusted analysis for any cluster characteristics that are imbalanced between the two study arms. Once the primary outcome is assessed, the investigators will likely use multivariate modeling to determine characteristics of women, in each study arm, who used any postpartum contraception within three months of delivery as compared to those who didn't, in both adjusted and unadjusted analysis. The plan is to use descriptive statistics to compare the other secondary outcomes between study arms (continuation and satisfaction). Finally, analysts will likely perform survival analysis of time to repeat pregnancy by study arm to observe if there is any statistically significant difference in the time to repeat pregnancy of women who became pregnant by twelve months in the study groups. In summary, our analysis plans a difference in differences analysis for our primary outcome, bivariate and multivariate analyses for our secondary outcome of any contraception use by study arm, descriptive statistics for our secondary outcomes of continuation and satisfaction rates among contraceptive users by study arm, and a survival analysis for time to repeat pregnancy by study arm.

ELIGIBILITY:
Inclusion Criteria:

* postpartum state
* enrolled in the Madres Sanas program
* able and willing to consent
* meeting age criteria
* not already received a contraceptive method

Exclusion Criteria:

* unable or unwilling to provide informed consent
* does not meet age criteria
* has already used a contraceptive method
* is pregnant

Ages: 15 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Postpartum state, which can only occur in females
Enrollment: 208 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2020-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margo S Harrison, MD, MPH, Principal Investigator — University of Colorado, Denver
Locations (2):
- University of Colorado, Aurora, Colorado, United States
- Fundacion para la Salud Integral de los Guatemaltecos, Caballo Blanco, Ritalhuleu, Guatemala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Harrison MS, Bunge-Montes S, Rivera C, Jimenez-Zambrano A, Heinrichs G, Bolanos A, Asturias E, Berman S, Sheeder J. Initial Contraceptive Choices of Women Enrolled in a Cluster-Randomized Trial in Southwest Trifinio, Guatemala. Matern Child Health J. 2022 Jan;26(1):168-176. doi: 10.1007/s10995-021-03275-4. Epub 2021 Oct 28. PMID 34709526
- [Derived] Harrison MS, Bunge-Montes S, Rivera C, Jimenez-Zambrano A, Heinrichs G, Bolanos A, Asturias E, Berman S, Sheeder J. Primary and secondary three-month outcomes of a cluster-randomized trial of home-based postpartum contraceptive delivery in southwest Trifinio, Guatemala. Reprod Health. 2020 Aug 20;17(1):127. doi: 10.1186/s12978-020-00974-z. PMID 32819394
- [Derived] Harrison MS, Bunge-Montes S, Rivera C, Jimenez-Zambrano A, Heinrichs G, Scarbro S, Juarez-Colunga E, Bolanos A, Asturias E, Berman S, Sheeder J. Delivery of home-based postpartum contraception in rural Guatemalan women: a cluster-randomized trial protocol. Trials. 2019 Nov 21;20(1):639. doi: 10.1186/s13063-019-3735-3. PMID 31752969

RESULTS

PARTICIPANT FLOW:
Groups:
- Postpartum Contraceptives Offered to Intervention Clusters: Participants were offered postpartum contraceptives (condoms, pills, injection, implant)
- Routine Care Offered to Control Clusters: Participants received routine counseling on postpartum contraception but did not have access to drugs and devices
Period: Overall Study
Arm/Group | Postpartum Contraceptives Offered to Intervention Clusters | Routine Care Offered to Control Clusters
Started | 108 (10/23/18) | 100 (10/23/18)
Completed (Primary Outcome Three Months) | 101 | 100
Not Completed | 7 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Postpartum Contraceptives Offered to Intervention Clusters | Routine Care Offered to Control Clusters | Total
Number analyzed (Participants) | 108 | 100 | 208
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 21.9 [18.8 to 25.4] | 21.8 [18.7 to 25.5] | 21.8 [18.7 to 25.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 100 | 208
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 108 | 100 | 208
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 108 | 100 | 208

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Implant Use at Three Months
Time Frame: Three months
Measure: Count of Participants; unit: Participants
Groups:
- Postpartum Contraceptives Offered to Intervention Clusters: offered pills, condoms, injectable, implant
- Routine Care Offered to Control Clusters: given contraceptive counseling
Arm/Group | Postpartum Contraceptives Offered to Intervention Clusters | Routine Care Offered to Control Clusters
Number analyzed (Participants) | 101 | 100
Participants | 28 | 2

2. Secondary Outcome: Number of Participants With Any Contraceptive Use at Three Months
Description: Participants actively using any contraceptive method three months after enrollment in the study as assessed by the three-month survey
Time Frame: 3 Months
Measure: Count of Participants; unit: Participants
Groups:
- Postpartum Contraceptives Offered to Intervention Clusters: patients opted for pills, condoms, injectable, or implant
- Routine Care Offered to Control Clusters: patients opted for a contraceptive method
Arm/Group | Postpartum Contraceptives Offered to Intervention Clusters | Routine Care Offered to Control Clusters
Number analyzed (Participants) | 101 | 100
Participants | 83 | 56

3. Secondary Outcome: Contraceptive Satisfaction at Twelve Months
Description: Participant satisfaction with any contraceptive method the woman might be using as determined by a survey question that asks if the woman is very satisfied, satisfied, dissatisfied, or very dissatisfied.
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Postpartum Contraceptives Offered to Intervention Clusters | Routine Care Offered to Control Clusters
Number analyzed (Participants) | 94 | 91
Participants
  "Very Satisfied" or "Satisfied" | 68 | 57
  "Dissatisfied" or "Very Dissatisfied" | 26 | 34

4. Secondary Outcome: Number of Participants With Contraceptive Continuation at Twelve Months
Description: Continuation of any contraceptive method a woman started in the postpartum period assessed by a survey at three and twelve months after study enrollment
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Postpartum Contraceptives Offered to Intervention Clusters | Routine Care Offered to Control Clusters
Number analyzed (Participants) | 94 | 91
Participants | 73 | 59

5. Secondary Outcome: Number of Participants With Repeat Pregnancy at Twelve Months
Description: Repeat pregnancy after enrollment in the study, as assessed at the enrollment (baseline) visit and at three and twelve months after study enrollment.
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Postpartum Contraceptives Offered to Intervention Clusters | Routine Care Offered to Control Clusters
Number analyzed (Participants) | 94 | 91
Participants | 0 | 4

ADVERSE EVENTS:
Time Frame: 16 months
Groups:
- Postpartum Contraceptives Offered to Intervention Clusters: pills, condoms, injectable, implant offerred
- Routine Care Offered to Control Clusters: contraceptive counseling given
Arm/Group | Postpartum Contraceptives Offered to Intervention Clusters | Routine Care Offered to Control Clusters
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/100
Other Adverse Events (participants affected / at risk) | 0/101 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-30): https://cdn.clinicaltrials.gov/large-docs/91/NCT04005391/Prot_SAP_000.pdf